CLINICAL TRIAL: NCT02665247
Title: Impact of Sleep Workshops in College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-00847
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Sleep; Insomnia; Sleep Deprivation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-SIP (Experimental): Participants assigned to the C-SIP group will attend sessions where information about sleep is presented. In session I, information about sleep and the effects of lack of sleep will be presented. Participants will also be presented with advice and tips on how to improve sleep. Session II will focus on assisting participants overcome any barriers they faced in applying the advice they received in session I; participants will also receive additional information on sleep and sleep-related techniques.
  Interventions: Behavioral: C-SIP
- Control Session (Other): Participants assigned to the control group will attend sessions in which information on sleep is presented in the form of dream discussions.
  Interventions: Other: Dream discussion

INTERVENTIONS:
Behavioral: C-SIP — In session I, information about sleep and the effects of lack of sleep will be presented. Participants will also be presented with advice and tips on how to improve sleep. Session II will focus on assisting participants overcome any barriers they faced in applying the advice they received in session I; participants will also receive additional information on sleep and sleep-related techniques.
  Arms: C-SIP
Other: Dream discussion — Participants assigned to the control group will attend sessions in which information on sleep is presented in the form of dream discussions.
  Arms: Control Session

SUMMARY:
The purpose of this pilot study is to assess the impact of sleep workshops on sleep, mood, anxiety and well-being measures in a sample of college students. College students have a high prevalence of sleep problems including poor sleep hygiene, volitional sleep deprivation, and insomnia. Sleep disorders in college students negatively affect mood, social functioning, physical safety, and academic performance. Rarely recognized by the students themselves, these conditions are therefore often untreated. Participants in this study will be randomly assigned to receive the College Sleep Improvement Plan (C-SIP) or a control session. Participants will be asked to track their sleep as well as complete questionnaires; a subset of participants will be asked to wear an activity monitor.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in classes at the NYU Washington Square campus

Exclusion Criteria:

* Students previously enrolled in the "While You Were Sleeping" course at NYU

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2019-11-24 (Actual); Study Completion 2019-11-24 (Actual)

PRIMARY OUTCOMES:
Change in Center for Epidemiologic Studies Depression Scale (CESD) score from baseline | 13 weeks
Change in Epworth Sleepiness Scale (ESS) score from baseline | 13 weeks
Change in Fatigue Severity Scale (FSS) score from baseline | 13 weeks
Change in Health Behaviors Survey (HBS) score from baseline | 13 weeks
Change in Morningness-Eveningness Questionnaire (MEQ-SA) from baseline | 13 weeks
Change in Perceived Stress Scale (PSS) score from baseline | 13 weeks
Change in Pittsburgh Sleep Quality Index (PSQI) score from baseline | 13 weeks
Change in Sleep Hygiene Index (SHI) score from baseline | 13 weeks
Change in State Trait Anxiety Inventory for Adults (Y-6 item) (STAI-Y6) score from baseline | 13 weeks
Change in Sleep Student Behavior Survey (SSBS) score from baseline | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jess Shatkin, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU School of Medicine, New York, New York, United States